CLINICAL TRIAL: NCT01754454
Title: Open-Label, Single-Center, Self Control, Phase Ⅰ/Ⅱ Clinical Trial to Evaluate the Safety and the Efficacy of Umbilical Cord-derived Mesenchymal Stem Cells in Patients With Acute Graft-versus-host Disease
Brief Title: Safety and Efficacy of UC-MSC in Patients With Acute Severe Graft-versus-host Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-CTC-MSC-002
Record Dates: First submitted 2012-11-11; First posted 2012-12-21 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-02

CONDITIONS: Acute GVH Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Human Umbilical Cord Derived MSC (Experimental): Human Umbilical Cord Derived MSC:
  Patients who receive standard of care plus treatment with ex vivo cultured adult human Umbilical Cord Derived Mesenchymal Stem Cells
  Interventions: Biological: Human Umbilical Cord Derived MSC

INTERVENTIONS:
Biological: Human Umbilical Cord Derived MSC — 1×10^6 UC-MSCs per kg intravenous injection the number of infusions: once a week, for four weeks in a row Time interval: estimate the condition of follow-up visit afer 28 days
  Other Names: UC-MSC

SUMMARY:
Allogenic haemopoietic stem cell transplantation (allo-HSCT) is the treatment for many malignant and non-malignant hematologic disorders. Acute graft-versus-host disease (aGVHD) is a serious life-threatening complication after allo-HSCT. The outcome for patients with aGVHD is poor and overall survival is low. Acute graft-versus-host disease (GVHD), as the major complication of allogeneic peripheral blood stem cell transplantation(PBSCT), limits the application of this curative therapy. Mesenchymal stem cells (MSCs) are multipotent stem cells, which are able to modulate immune response in vitro and in vivo, and have possibilities of treating diseases caused by immune dysregulation such as aGVHD. MSCs obtained from umbilical cord (UC) have similar immunosuppressive properties as bone marrow-MSCs. In addition, UC-derived MSCs can be used for off-the-shelf use and are obtained without any harm to donors than bone marrow-MSCs. Therefore, the investigators designed this study to evaluate the safety and efficacy of UC-derived MSCs in patients with aGVHD.

DETAILED DESCRIPTION:
The mesenchymal stem cells (MSC) is a class of low immunogenicity from mesoderm, had the self-renewal and differentiation potential as pluripotent stem cells. The umbilical cord is one of the important sources of MSC. Human UC-MSC compared with the bone marrow-derived MSC has the following advantages: (1) the umbilical cord, as a "waste" after giving birth can be obtained without any harm to the donor. (2) easy available, and no ethical issues. (3) its likelihood of contamination is small because of the protection of the placental barrier. (4) human UC-MSC has a stronger amplification capacity, a shorter doubling time, a higher colony forming efficiency and lower immunogenicity. (5) which avoids the activity and differentiation of bone marrow-derived MSC latent with the donor disadvantage of increasing age decreased.

human UC-MSC not only for hematopoietic stem cell graft implantation and amplification has a role in promoting and exhibit immunomodulatory effects and characteristics of damaged or targeted sites of chronic inflammation. human UC-MSC in the prevention and treatment of graft-versus-host disease (GVHD) induced organ transplantation immune tolerance and other fields has broad application prospects.

After more than 10 years of exploration, the investigators and other practitioners caught studies found that the umbilical cord is more suitable as mesenchymal stem cells seed cells relative to the bone marrow, umbilical cord easily obtained, no ethical issues, better amplification ability in vitro, viral contamination risk is small, and many other advantages. Therefore, over the years, the investigator team for the umbilical cord mesenchymal stem cells in a lot of the basic work has been confirmed that mesenchymal stem cells derived from the umbilical cord had safety and effectiveness in in the treatment of acute graft versus host disease in zoology test, and successfully establish a perfect umbilical cord mesenchymal stem cells in standard operating procedures (including screening umbilical cord, large-scale preparation, quality inspection, preservation, recovery, transportation, infusion, etc.). The investigators will carry out the clinical research based on above preliminary results.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70 years
* undergoing allogeneic hematopoietic stem cell transplant recipients
* post-transplant acute GVHD (Ⅲ ~ Ⅳ degrees)
* the effects of other immunosuppressive therapy
* glucocorticoid resistance or glucocorticoid therapy invalid
* cooperation observed adverse events and efficacy
* patients understand the status of the experimental observations, with the doctor's treatment and post-treatment follow-up, patients or their legal representatives signed a written informed consent

Exclusion Criteria:

* had severe allergy history
* within three months to participate in other medical or drug trials
* as a subjects was sampled within three months
* smoking, alcohol and drug abusers
* suffers from an important organ of primary disease (heart, liver, kidney, lung, brain, etc.), infectious diseases (including HIV and suspicious latent infection), people with disabilities and / or mental disorders
* to judge according to the researchers, the subjects could not complete the study or may not be able to comply with the requirements of this study (due to administrative reasons or other reasons)

Exit criteria:

* In clinical trials, the participants had some complications, complications or special physiological changes, unfit to continue to accept the test
* subjects with poor compliance, affect the determination of the pharmacokinetic results
* subjects using the drugs may affect the results of the pharmacokinetic
* the occurrence of serious adverse events in subjects
* subjects withdrew informed consent, or withdraw from the trial itself

Termination criteria:

* serious adverse events (except the researchers judgment and research drugs must be independent), should stop all test
* found that clinical research plan has important lapses, difficult to evaluate the effects of drugs, or a better design in implementation had an important deviation, difficult to continue to evaluate the effects of drugs
* sponsor for the request to terminate (such as funds reason, management reason, etc.)
* state food and drug administration for some reason ordered to terminate test

Exclusion criteria:

* does not meet the entry criteria
* exclusion criteria
* once the drug is not used in
* no records

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Safety of UC-MSC in patients with acute graft-versus-host disease | 180 days
  * vital signs
  * adverse events related to infusion
  * physical examination indexes
  * Eastern Cooperative Oncology Group(ECOG)performance status
  * mixed lymphocyte reaction(MLR)

SECONDARY OUTCOMES:
Efficacy of UC-MSC in patients with acute graft-versus-host disease | 180 days
  * Complete, partial response rate at 28 and 180 days
  * Complete response(CR)rate (%)=(number of CR/number of participants)*100%
  * Partial response(PR)rate (%)=(number of PR/number of participants)*100%

CONTACTS AND LOCATIONS:
Overall Officials: Hu Chen, M.D., Ph.D., Study Chair — Department of Hematopoietic Stem Cell Transplantation, Affiliated Hospital to Academy of Military Medical Sciences; Bin Zhang, M.D. Ph.D, Study Director — Department of Hematopoietic Stem Cell Transplantation, Affiliated Hospital to Academy of Military Medical Sciences
Locations (2):
- China (2):
  - Department of Hematopoietic Stem Cell Transplantation, Beijing
  - Department of Hematopoietic Stem Cell Transplantation, Affiliated Hospital to Academy of Military Medical Sciences, Beijing

REFERENCES:
- [Derived] Niu JW, Li Y, Xu C, Sheng H, Tian C, Ning H, Hu J, Chen J, Li B, Wang J, Lou X, Liu N, Su Y, Sun Y, Qiao Z, Wang L, Zhang Y, Lan S, Xie J, Ren J, Peng B, Wang S, Shi Y, Zhao L, Zhang Y, Chen H, Zhang B, Hu L. Human umbilical cord-derived mesenchymal stromal cells for the treatment of steroid refractory grades III-IV acute graft-versus-host disease with long-term follow-up. Front Immunol. 2024 Aug 15;15:1436653. doi: 10.3389/fimmu.2024.1436653. eCollection 2024. PMID 39211037